CLINICAL TRIAL: NCT06333236
Title: Effect of Kron (Citicoline and Nicotinamide Oral Solution) on Patients With Open-angle Glaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ASST Santi Paolo e Carlo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OCU_KRON
Record Dates: First submitted 2024-02-01; First posted 2024-03-27 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Food

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group KRON (Experimental): Active Treatment: Kron® (300ml) oral solution containing citicoline free acid 40 mg/ml; nicotinamide 15 mg/ml. In addition to the IOP-lowering medications, Kron will be administered at a dosage of 10 ml in the morning. To each patient will be given two bottles during the baseline visit and will be asked to return them at the end of the study (3 month) for the compliance assessment.
  Interventions: Other: Food for Special Medical Purposes: Kron®
- Control Group (No Intervention): No interviention in addition to the IOP-lowering medications.

INTERVENTIONS:
Other: Food for Special Medical Purposes: Kron® — Citicoline 40mg/ml + Nicotinamide 15 mg/ml oral solution
  Arms: Group KRON

SUMMARY:
Aim of this study is to investigate the administration effects of the combination of citicoline 40mg/ml and nicotinamide 15mg/ml oral solution (Kron®) on short term improvement in inner retinal function, bioelectrical activity of the visual cortex and visual function.

DETAILED DESCRIPTION:
Prospective, masked, randomized placebo-controlled study to evalute the offect of the oral solution Kron® (citicoline 40mg/ml and nicotinamide 15mg/ml) on patients with a diagnosis of open angle glaucoma and risk of glaucoma progression.

Glaucomatous patients with a diagnosis of open angle glaucoma and risk of glaucoma progression who meet the study criteria will be enrolled and randomly assign to the following two arms:

1. Treatment group (TG): 20 patients will receive Citicoline 40 mg/ml + Nicotinamide 15 mg/ml oral solution for 3 months (10 ml/day)
2. Control group (CG): 10 patients will be evaluated as control

Once recruited, a clinical evaluator will perform a comprehensive ophthalmologic evaluation at baseline, week 6 and week 12. The following examinations will be done in the following sequence:

* Visual acuity
* Slit lamp evaluation
* PERG
* PEV pattern
* Tonometry
* Visual field
* Optical Coherence Tomography
* Dilated Fundus examination

ELIGIBILITY:
Inclusion Criteria:

* glaucomatous patients with moderate visual field loss, MD ranging from -6 dB and -12 dB, and risk of progression
* controlled intraocular pressure
* at least 3 previous visual field examinations.

Exclusion Criteria:

* angle closure glaucoma and secondary open angle glaucoma
* refractive error outside +2D and -6D
* ophthalmic surgery 6 months before the recruitment
* presence of cataract or other conditions that could affect results of perimetry or electroretinography
* treatment with supplements in any form with a demonstrated or presumed neuroprotecting/neuroenhancing effect in the last six months
* presence of other ocular or systemic diseases that could affect results of perimetry or electroretinography.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-04-10 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-09-14 (Actual)

PRIMARY OUTCOMES:
Electrofunctional evaluation | 3 months
  Short term improvement in inner retinal function and bioelectrical activity of the visual cortex evaluated by means of PERG (P50 and N95 peaks) and PEV (P100 implicit time and N75-P100 amplitude) pattern.

SECONDARY OUTCOMES:
VF and SD-OCT | 3 months
  Visual field examination will be performed at the beginning and at the end of trial. Standard pattern short-term improvement in visual function in treated patients evaluated by means of VF. Retinal nerve fiber layer thickness, ganglion cell complex thickness and minimum rim width will be evaluated at the baseline and at the end of the study.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - ASST Santi Paolo e Carlo, Milan, Mi
  - Luca Rossetti, Milan, MI